CLINICAL TRIAL: NCT03931993
Title: A Pre-Season,Randomized,Single-blind,Placebo-controlled,Parallel-group Study to Determine Tolerability+Safety of a New Cumulative Dose of GrassMATAMPL Compared With Placebo in Patients With Seasonal Allergic Rhinoconjunctivitis Due to Grass Pollen Allergy
Brief Title: A Study of Tolerability and Safety of a New Cumulative Dose of Grass MATA MPL
Acronym: G104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Collaborators: SynteractHCR (Industry); Metronomia Clinical Research GMBH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GrassMATAMPL104
Record Dates: First submitted 2017-03-29; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Grass MATA MPL; Safety
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Intervention Model Description: Single-blind
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1 (Placebo Comparator): Six 1.0mL placebo injections (2% w/v L-tyrosine)
  Interventions: Biological: Placebo comparator
- Treatment Group 2 (Experimental): Six 1.0mL injections of Grass MATA MPL 900, 2700, 8000, 8000, 8000, and 8000 SU
  Interventions: Biological: Grass MATA MPL

INTERVENTIONS:
Biological: Placebo comparator
  Arms: Treatment Group 1
Biological: Grass MATA MPL
  Arms: Treatment Group 2

SUMMARY:
There is increasing evidence that the effectiveness of allergy immunotherapy to control symptoms of rhinoconjunctivitis is related to the cumulative dose of allergen or allergoid administered during a single regimen of subcutaneous (SC) injections or of sublingual administration. Previously, high cumulative doses of the Grass MATA MPL 10200 and 18200 SU (Standardized Units) were compared with the marketed dose of 5100 SU and were found to have acceptable tolerability and safety. The purpose of this study is to evaluate the tolerability and safety of an even higher cumulative dose regimen of 35600 SU. of Grass MATA MPL compared with placebo in patients with seasonal allergic rhinoconjunctivitis (SAR) due to grass pollen, to enable selection of the best dose to take forward for further development.

DETAILED DESCRIPTION:
This will be a placebo-controlled study, using a 1:1 randomization and parallel-group, single-blind design, in patients with seasonal allergic rhino-conjunctivitis to grass pollen conducted at multiple centres in the US. The study will be conducted outside the grass pollen season and is comprised of 3 periods.

* Period 1: Screening
* Period 2: Randomization and treatment
* Period 3: Post-treatment safety follow-up

Period 1 consists of the screening visit (Visit 1) at which patient eligibility will be assessed. Blood samples will be taken for clinical safety laboratory assessments and for baseline transcriptomics analysis. Eligible patients will proceed to Period 2 for enrolment into study.

Period 2 starts with the randomization visit (Visit 2: 3-33 days after Visit 1), at which eligible patients will be randomly allocated to the Grass MATA MPL 35600 SU or placebo treatment groups and receive the first of 6 weekly injections of subcutaneous immunotherapy (SCIT). Injections 2 to 6 will be administered at Visits 3 to 7. After each injection, patients will be kept under observation at the site for at least 30 minutes by personnel qualified to observe for and manage local and systemic adverse events. This period may be extended by the investigator according to his/her judgment. The observation will be followed up by a telephone call approximately 24 hours after the time of injection. In the event of mild or moderate systemic adverse events judged by the investigator to be well-tolerated by the patient and to show good recovery, the patient may continue treatment as scheduled.

Period 3 (Visit 8 - End of Study) will occur 6-8 days after Visit 7 to review any AEs and to perform end-of-treatment assessments, which will include blood draws for safety laboratory tests and transcriptomics analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a positive skin prick test for grass pollen allergen.
* Positive skin prick test to positive histamine control
* Negative skin prick test to negative control
* Specific IgE for grass pollen as documented by ImmunoCAP test with class ≥ 2
* A history of moderate to severe symptoms of seasonal allergic rhinitis and/or conjunctivitis due to grass (Pooideae) pollen exposure that required repeated use of antihistamines, nasal steroids, and/or leukotriene modifiers for relief of symptoms during the last two consecutive seasons prior to the study
* Males or non-pregnant, non-lactating females who are not of child-bearing potential or using effective contraception
* Patients who are normally active and otherwise judged to be in good health
* For patients with a history of asthma, forced expiratory volume in 1 second (FEV1) ≥ 80% of National Health and Nutrition Examination Surveys (NHANES) predicted, with a FEV1/forced vital capacity (FVC) ratio ≥ 70%.
* Able to observe the drug washout times listed in the Prohibited Medications Table below prior to screening
* Patients willing and able to attend required study visits and able to follow the protocol requirements.
* Patients willing and able to give written informed consent.

Exclusion Criteria:

* Symptoms outside the grass pollen season due to a perennial and/or non-grass seasonal allergen, if the patient is unable to avoid the offending allergen.
* Immunological disorders or other diseases that in the opinion of the investigator may pose a safety risk.
* Presence of moderate to severe asthma, characterized by the current use of inhaled steroids at a daily dose above 400 micrograms of budesonide (or equivalent)
* Emergency room visit or admission for asthma in the 12 months prior to Visit 1 or history of a life-threatening asthma attack ever.
* Presence of non-atopic rhinitis and/or rhino-sinusitis (with or without polyps).
* Presence of any skin conditions (skin abnormalities, tattoos etc.) which might interfere with the interpretation of the SPT results.
* Current diagnosis of type I diabetes. Patients with type II diabetes will only be allowed to participate at the discretion of the investigator.
* Treatment with a preparation containing MPL (e.g. Cervarix) within 6 months prior to screening
* Moderate to severe upper or lower respiratory tract infections requiring medication within 14 days of or a diagnosis of sinusitis within 30 days of randomisation
* Clinical history of severe or life-threatening anaphylactic reactions to foods, insect venom, exercise, drugs or idiopathic anaphylaxis.
* Clinical history of allergy, hypersensitivity or intolerance to the excipients of the study medication.
* Tyrosine metabolism disorders, especially tyrosinemia and alkaptonuria.
* Unable to receive epinephrine therapy (i.e., use of epinephrine is contraindicated).
* Clinical history of immunodeficiency, including those who are on immunosuppressant therapy.
* Clinical history of recurrent idiopathic angioedema.
* Beta-blocker medication, including eye drops, for any indication.
* Treatment with monoamine oxidase inhibitors, tricyclic antidepressants or ACE inhibitors.
* Clinical history of drug or alcohol abuse which, in the investigator's opinion, could interfere with the patient's ability to participate in the study.
* Participation in a clinical research trial with any investigational medicinal product within 4 weeks of screening or concomitantly with this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Number and frequency of adverse events (AEs) | 36 - 48 days
Number and frequency of adverse reaction complexes (ARCs) | 36 - 48 days
  The maximum intensity of all injection site [local] and systemic AEs experienced by a patient within a 24-hour period after an injection.
Frequency of premature discontinuation from treatment or study due to AEs. | 36 - 48 days
Changes in vital sign parameters at all visits in the treatment period from pre-injection to post-injection - Systolic blood pressure | 30 - 40 days
  Mean values compared to normal range
Changes in vital sign parameters at all visits in the treatment period from pre-injection to post-injection - Diastolic blood pressure | 30 - 40 days
  Mean values compared to normal range
Changes in vital sign parameters at all visits in the treatment period from pre-injection to post-injection - Pulse | 30 - 40 days
  Mean values compared to normal range
Changes in vital sign parameters at all visits in the treatment period from pre-injection to post-injection - Body temperature | 30 - 40 days
  Mean values compared to normal range
Changes in routine clinical laboratory values - Serum Chemistry | 36 - 48 days
  Absolute and relative number of patients with values below, within or above the normal range
Changes in routine clinical laboratory values - Hematology | 36 - 48 days
  Absolute and relative number of patients with values below, within or above the normal range
Changes in routine clinical laboratory values - Urinalysis | 36 - 48 days
  Absolute and relative number of patients with values below, within or above the normal range
Changes in peak expiratory flow rate (PEFR) before and after injections in asthmatic patients | 30 - 40 days

SECONDARY OUTCOMES:
Number and frequency of neuro-inflammatory (NI) events. | 36 - 48 days
  Assessed by clinical judgement
Number and frequency of new onset autoimmune disease (NOAD) events. | 36 - 48 days
  Assessed by clinical judgement

OTHER OUTCOMES:
Transcriptomics analysis | 36-48 days
  X fold-change in expression of selected genes (before and after the treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Higenbottam, MD, FRCP, Study Director — Allergy Therapeutics
Locations (4):
- United States (4):
  - Vedas Research, Edison, New Jersey
  - Atlantic Reseach Center, Ocean City, New Jersey
  - STARx Asthma and Allergy Center, Springfield, New Jersey
  - Allergy Partners of New Jersey, Teaneck, New Jersey

IPD SHARING:
Plan to Share IPD: No